CLINICAL TRIAL: NCT06703099
Title: Effects of Magnesium Supplementation on Body Composition in Physically Active Individuals: A Pilot Study
Brief Title: Magnesium Supplementation on Body Composition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: Life Extension Foundation Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-432-NSU
Record Dates: First submitted 2024-11-10; First posted 2024-11-25 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Body Composition Changes
Keywords: body composition; magnesium; lean body mass; InBody; Active; Pilot study
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnesium Supplementation (Experimental): Life Extension® Extend Release Magnesium 250 mg/day of oral magnesium in capsule form to be taken once a day at breakfast/morning.
  Interventions: Dietary Supplement: Magnesium Supplementation

INTERVENTIONS:
Dietary Supplement: Magnesium Supplementation — Life Extension® Extend Release Magnesium 250 mg/day of oral magnesium in capsule form to be taken once a day at breakfast/morning over 8 weeks.

SUMMARY:
The goal of this interventional clinical trial is to learn if the supplementation of magnesium can affect body composition in physically active individuals between the ages of 18 and 30. The main question[s] it aims to answer [is/are]:

How does magnesium supplementation affect body composition in physically active individuals?

Participants will take a magnesium capsule once daily for 8 weeks, log their food intake into MyFitnessPal 3 days weekly for the 8 weeks, keep their physical activity consistent to their current regimen, and have 1 baseline appointment with 2 follow ups evenly dispersed (mid-point and post-intervention).

DETAILED DESCRIPTION:
This study's research design is a pilot single-arm intervention trial. Data collection will occur three times (baseline, midpoint, and post-intervention) over the course of the 8 week intervention period. Data collection will take place on Nova Southeastern University Campus (3301 S University Dr, Davie, FL 33328). Eligible participants will undergo an 8-week supplementation regimen with Life Extension® Extend Release Magnesium, containing a 250 mg/capsule blend of ZümXR® magnesium oxide and magnesium citrate. The supplement will be distributed to participants at baseline and midpoint measurement assessments. Dietary intake will be monitored at least 3 days of the week for the 8 week intervention period using the MyFitnessPal app. Participants will be instructed not to change their eating habits for the duration of the intervention. Outside of their usual physical activity training, participants will be instructed not to change their physical activity habits for the duration of the intervention. Body composition will be assessed at baseline, midpoint, and post-intervention using Bioelectrical Impedance Analysis (BIA). Participants will be instructed to wear light clothing (with no zippers, belts, or buttons), remove all jewelry before testing, not consume any food 3-4 hours before testing, not drink caffeine on the day of testing, and hydrate adequately prior to testing. Demographic information (age, sex, and physical activity status) will be assessed via a simple questionnaire at baseline.

Order of events:

* Distribute recruitment through flyers at NSU Main Campus (Davie).
* Screening process via demographic survey to determine qualification based on participant inclusion/exclusion criteria.Sign consent forms, explain procedures and study outcomes to participants.
* Baseline anthropometric measurements (Bioelectrical Impedance Analysis (BIA) [InBody 270; InBody Co., Ltd. (Seoul, Korea)], height, and weight) and diet analysis (MyFitnessPal Nutrition Tracking App).
* Distribute supplements for the first 4 weeks of intervention (Life Extension Extend Release Magnesium, 28 capsules/participant).
* Bi-weekly follow ups with participants via phone (2 follow ups).
* Midpoint anthropometric measurements (BIA [InBody 270; InBody Co., Ltd. (Seoul, Korea)] and diet analysis (MyFitnessPal Nutrition Tracking App). Perform capsule counting.
* Distribute supplements for the last 4 weeks of intervention (Life Extension Magnesium Caps, 28 capsules/participant).
* Bi-weekly follow ups with participants via phone (2 follow ups).
* Final anthropometric measurements (BIA [InBody 270; InBody Co., Ltd. (Seoul, Korea)] and diet analysis (MyFitnessPal Nutrition Tracking App). Perform capsule counting.

Data collection:

Height and weight will be collected at baseline, midpoint, and post-intervention visits using weight scale and stadiometer. BMI will be calculated using height and weight. Body composition will be assessed using a multi-frequency Bioelectrical Impedance Analysis (BIA) device [InBody 270; InBody Co., Ltd. (Seoul, Korea)].

Participants will be required to keep a food diary for at least 3 days per week using the MyFitnessPal (MFP) Nutrition Tracking Smartphone Application. Similar software has been shown to produce results comparable to other, more time-intensive methods of dietary data collection such as 24-hour recalls. Participants' diets will be analyzed during the baseline and midpoint assessment visits using the MyFitnessPal (MFP) Nutrition Tracking App. Diet analyses will be conducted to determine how much dietary magnesium and protein participants are consuming in their normal diet, as both factors may affect LBM accrual.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years old
* classified as a physically active individual for at least 1 year defined as being any individual that regularly engages in the minimum physical activity requirements as put forth by the American College of Sports Medicine.
* have a BMI of 19-30 kg/m2

Exclusion Criteria:

* smokers
* have been diagnosed with any metabolic/chronic disease
* are taking medications that can interfere with body composition
* are unwilling to follow study guidelines
* have a current physical condition that may be exacerbated by physical activity as determined by their general practitioner
* are pregnant or intend to become pregnant within 3 months
* have taken Mg supplements within the last 6 months
* are using steroids or any anabolic agents
* have pacemakers, implants, or any non-removable metal surgical implants

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-04-27 (Actual)

PRIMARY OUTCOMES:
Body Composition - BMI | 8 weeks
  Using the InBody 270, height and weight will be combined to report BMI (kg/m2)
Body Composition - Weight | 8 weeks
  Using the InBody 270, weight will be reported in pounds (lb)
Body Composition - LBM | 8 weeks
  Using the InBody 270, lean body mass (LBM) will be reported in pounds (lb)
Body Composition - BFM | 8 weeks
  Using the InBody 270, body fat mass (BFM) will be reported in pounds (lb)

SECONDARY OUTCOMES:
Dietary Intake | 8 weeks
  Dietary intake inclusive of Mg (in milligrams) in food items and total protein (in grams) using Food Logs

CONTACTS AND LOCATIONS:
Overall Officials: Madison M Doten, BS, Principal Investigator
Locations (1):
- Nova Southeastern University HPD Annex Building, Davie, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Statistical analysis of data will be shared, however individual documentation for participants will be kept on file and destroyed after 36 months as per IRB protocol. These documents will not be available to other researchers.

DOCUMENTS (1):
  • Informed Consent Form (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT06703099/ICF_000.pdf